CLINICAL TRIAL: NCT05144542
Title: The Potential Risks and Benefits of Electronic Cigarettes to Older Smokers at High Risk for Lung Cancer
Brief Title: Risk and Benefits of Electronic Cigarettes to Older Smokers at High Risk for Lung Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2019-1266; NCI-2021-03212 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-1266 (Other: M D Anderson Cancer Center); R01CA238478 (NIH)
Record Dates: First submitted 2021-11-18; First posted 2021-12-03 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Lung Carcinoma
MeSH Terms: conditions — Lung Neoplasms | interventions — Nicotine Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- E-Cigarettes (Experimental): Participants vape e-cigarettes for 26 weeks. Participants use smartphone to answer questions about nicotine cravings and mood, and log daily smoking activity every day for up to 182 days. Participants complete questionnaires over 50 minutes and undergo collection of urine sample at 0, 1, 7, 13, and 27 weeks, and collection of blood samples at 6, 12, and 26 weeks. Participants may also undergo measurement of CO levels at 1, 6, 12, and 26 weeks.
  Interventions: Procedure: Participants smoke their usual brand of cigarettes for 26 weeks.; Procedure: Participants will vape electronic cigarettes for 26 weeks.; Drug: Nicotine Replacement; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Participants smoke their usual brand of cigarettes for 26 weeks. — Participants smoke their usual brand of cigarettes for 26 weeks.
Procedure: Participants will vape electronic cigarettes for 26 weeks. — Participants will vape electronic cigarettes for 26 weeks.
Drug: Nicotine Replacement — Smoke usual brand of cigarettes
  Other Names: Nicotine Replacement Therapy; NRT
Drug: Nicotine Replacement — Vape e-cigarettes
  Other Names: Nicotine Replacement Therapy; NRT
Other: Questionnaire Administration — Use smartphone to answer questions about nicotine cravings and mood, and log daily smoking activity every day.

SUMMARY:
This clinical trial investigates the effects of switching from smoking regular cigarettes to electronic cigarettes (e-cigarettes) among older adult smokers at high risk for lung cancer. E-cigarettes use heated vapor to deliver nicotine. Information gained from this trial may help inform regulators of the potential risks and benefits of switching smokers at high risk for lung cancer to electronic cigarettes. This research also may help inform the Food and Drug Administration (FDA) how best to regulate e-cigarettes with the goal of improving public health.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To characterize the effects of switching from combustible cigarettes (CCs) to e-cigarettes (ECs) on product use, product acceptability, and reinforcement among adult daily CC smokers at high risk for lung cancer.

SECONDARY OBJECTIVE:

I. To characterize the effects of switching from CCs to ECs on biomarkers of inflammation and oxidative stress among adult daily CC smokers at high for lung cancer.

EXPLORATORY OBJECTIVES:

I. To characterize metabolomic changes that result from switching from CCs to ECs among CC smokers at high risk for lung cancer.

II. To character which factors moderate or mediate the effects of switching from CCs to ECs among CC smokers at high risk for lung cancer.

Outline:

Participants are assigned to switch to e-cigarettes.

ELIGIBILITY:
Inclusion Criteria:

* Aged 50-80 years who currently smokes at least 1 or more combustible cigarettes per day OR who is a nondaily smoker (any self-reported smoking in the past 30 days) with a 20 pack-year history.
* Being interested in trying ECs to change CC smoking behavior
* Willing to have biospecimen samples taken, either in-home using a mobile phlebotomoty service, or at an approved collection site
* Have an address where he/she can receive mail
* Being fluent in spoken and written English
* Agrees to comply with all MD Anderson institutional policies related to COVID-19 screening prior to any in-person research visit.
* The individual agrees to not engage in study procedures or interactions with study personnel while operating a vehicle.

Exclusion Criteria:

* Individuals who report depressive symptoms in the moderately severe or severe range on the PHQ-9 (scores of 15 or above); or who report current suicidal ideation on the PHQ-9
* Have ever had a diagnosis of lung cancer, have uncontrolled or unstable medical condition (e.g., uncontrolled hypertension, angina, diabetes)
* Unwilling to consent for blood draw
* Evidence of cognitive deficits or instability that would preclude reliable study participation
* Being pregnant, engaging in breast-feeding, or being of childbearing potential and engaging in sexual activity that could lead to pregnancy and is not protected by a medically acceptable, effective method of birth control while enrolled in the study, as determined by self-report. Medically acceptable contraceptives include: (1) approved hormonal contraceptives (such as birth control pills, patches, implants or injections), (2) barrier methods (such as a condom or diaphragm) used with a spermicide, or (3) an intrauterine device (IUD). Contraceptive measures sold for emergency use after unprotected sex are not acceptable methods for routine use.
* Considered by the investigator to be an unsuitable or unstable candidate (including but not limited to the following situations: unwilling or unable to comply with study procedures)
* Individuals who reside in an area that is outside of our shipping company or mobile phlebotomty contractors' areas of operation or in a jurisdiction outside of our medical staff's licensure (if unable to attend in-person clinic visits) AND who decline to come in to clinic to provide necessary samples and/or collect study products.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-03-07 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Cigarettes per day | Up to 182 days
  Will be collected using smartphone daily diary data of combustible cigarette use over last 24 hours.

SECONDARY OUTCOMES:
High-sensitivity C-reactive protein (hs-CRP) | through study completion, an average of 1 year
  This measure will be collected using blood draws at weeks 0, 6, 12, and 26.
White blood cells (WBC) | through study completion, an average of 1 year
  This measure will be collected using blood draws at weeks 0, 6, 12, and 26.
8-epi prostaglandin F2 alpha (8-epi-PGF2a) | through study completion, an average of 1 year
  This measure will be collected using blood draws at weeks 0, 6, 12, and 26.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Robinson, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org